CLINICAL TRIAL: NCT03534986
Title: Effect of High Frequency Chest Wall Oscillation Vests on Spirometry Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Biophysics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02
Record Dates: First submitted 2018-05-14; First posted 2018-05-23 (Actual); Results first posted 2018-09-06 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Cystic Fibrosis; Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- AffloVest The Vest Arm (Experimental): Devices placed on highest intensity / highest frequency
  Interventions: Device: International Biophysics AffloVest; Device: Hill-Rom The Vest
- AffloVest inCourage Arm (Experimental): Devices placed on highest intensity / highest frequency
  Interventions: Device: International Biophysics AffloVest; Device: Respirtech inCourage
- AffloVest SmartVest Arm (Experimental): Devices placed on highest intensity / highest frequency
  Interventions: Device: International Biophysics AffloVest; Device: Electromed SmartVest

INTERVENTIONS:
Device: International Biophysics AffloVest — High-frequency chest wall oscillation vest
Device: Hill-Rom The Vest — High-frequency chest wall oscillation vest
  Arms: AffloVest The Vest Arm
Device: Respirtech inCourage — High-frequency chest wall oscillation vest
  Arms: AffloVest inCourage Arm
Device: Electromed SmartVest — High-frequency chest wall oscillation vest
  Arms: AffloVest SmartVest Arm

SUMMARY:
The impact of high-frequency chest wall oscillation therapy on spirometry values (Forced Expiratory Volume, Forced Vital Capacity, Peak Expiratory Flow, Forced Expiratory Flow and Tidal Volume is investigated during use of several products and comparing to baseline values.

DETAILED DESCRIPTION:
The study will be broken into three (3) arms:

* AffloVest® & The Vest®
* AffloVest® & inCourage®
* AffloVest® & SmartVest® Subjects will be randomly assigned to an arm. Within each arm, the order of products will be also randomized.

Baseline spirometry (Forced Expiratory Volume (FEV1), Forced Vital Capacity (FVC), Peak Expiratory Flow (PEF), Forced Expiratory Flow (FEF25-75%) and Tidal Volume (TV)) will be taken at the beginning, middle and end of each series of measurements with each subject, without any device on the subject.

A product (AffloVest or Compressor-based vest) will be placed onto subject and turned ON to the highest frequency and intensity settings. Then the subject will be given a certain period of time to adjust and spirometry measurements will then be repeated, then The product will be removed and the subject will be allowed a recovery period, then the other product will be placed on the subject, turned ON and spirometry measurements will repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject, ages 18 - 50

Exclusion Criteria:

* Non-ambulatory, diagnosed neuromuscular disorder, currently using any type of oscillation vest therapy, diagnosed co-morbid condition (i.e. lung cancer, other lung disorder or disease), currently enrolled in a medical research study, non-English speaking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W O'Brien, MD, Principal Investigator — PDS Research
Locations (1):
- PDS Research, Kissimmee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AffloVest The Vest Arm | AffloVest inCourage Arm | AffloVest SmartVest Arm
Started | 10 | 10 | 12
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AffloVest The Vest Arm | AffloVest inCourage Arm | AffloVest SmartVest Arm | Total
Number analyzed (Participants) | 10 | 10 | 12 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 12 | 32
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (11.9) | 30.6 (13.3) | 34.7 (10.2) | 31.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 7 | 13
  Male | 8 | 6 | 5 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: TV
Description: Tidal Volume, the lung volume representing the normal volume of air displaced between normal inhalation and exhalation when extra effort is not applied
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L
Groups:
- Baseline: Patient Baseline Results
- AffloVest Arm: Devices placed on highest intensity / highest frequency
  Hill-Rom The Vest: High-frequency chest wall oscillation vest
- Compressor Arm: Devices placed on highest intensity / highest frequency
  Compressor-type device
Arm/Group | Baseline | AffloVest Arm | Compressor Arm
Number analyzed (Participants) | 10 | 10 | 10
L | 0.93 [0.30 to 2.32] | 1.00 [0.27 to 2.28] | 1.07 [0.24 to 2.69]

2. Primary Outcome: PEF
Description: Peak Expiratory Flow, a person's maximum speed of expiration
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L/s
Arm/Group | Baseline | AffloVest Arm | Compressor Arm
Number analyzed (Participants) | 10 | 10 | 10
L/s | 8.19 [3.96 to 11.82] | 8.28 [3.50 to 12.00] | 8.13 [4.23 to 12.89]

3. Primary Outcome: FVC
Description: Forced Vital Capacity, the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L
Arm/Group | Baseline | AffloVest Arm | Compressor Arm
Number analyzed (Participants) | 10 | 10 | 10
L | 4.29 [2.48 to 6.57] | 4.25 [2.5 to 7.42] | 4.12 [2.29 to 6.73]

4. Primary Outcome: FEV1
Description: Forced Expiratory Volume, the volume of air that can be forced out in one second after taking a deep breath
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L
Arm/Group | Baseline | AffloVest Arm | Compressor Arm
Number analyzed (Participants) | 10 | 10 | 10
L | 3.51 [2.05 to 5.54] | 3.46 [2.00 to 6.19] | 3.30 [1.92 to 5.83]

5. Primary Outcome: FEF25-75%
Description: Forced Expiratory Flow (25-75%), the peak expiratory flow at 25 - 75% FVC
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L/s
Arm/Group | Baseline | AffloVest Arm | Compressor Arm
Number analyzed (Participants) | 10 | 10 | 10
L/s | 3.71 [1.77 to 6.43] | 3.54 [1.63 to 6.37] | 3.19 [1.19 to 6.22]

ADVERSE EVENTS:
Time Frame: Study enrollment, approximately 2 hours.
Arm/Group | AffloVest The Vest Arm | AffloVest inCourage Arm | AffloVest SmartVest Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03534986/Prot_SAP_000.pdf